CLINICAL TRIAL: NCT01015170
Title: The STOP Study: Real World Effectiveness of Zyban Treatment in a Clinical Population
Brief Title: STOP Study: Effectiveness of Zyban in a Clinical Population
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government)
Responsible Party: Principal Investigator, Dr. Peter Selby, Clinician Scientist, Addictions Program, Centre for Addiction and Mental Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 005/2008
Record Dates: First submitted 2009-11-17; First posted 2009-11-18 (Estimated); Results first posted 2017-03-27 (Actual); Last update posted 2017-03-27 (Actual); Status verified 2017-02

CONDITIONS: Cigarette Smoking; Nicotine Addiction; Smoking Cessation
Keywords: smoking cessation; nicotine addiction; Zyban; bupropion hydrochloride
MeSH Terms: conditions — Cigarette Smoking; Tobacco Use Disorder; Smoking Cessation | interventions — Bupropion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bupropion HCl (Experimental): Up to 8 week of bupropion SR (150mg BID) + counseling.
  Interventions: Drug: bupropion HCl

INTERVENTIONS:
Drug: bupropion HCl — 150mg BID for up to 8 weeks + counseling
  Other Names: Zyban

SUMMARY:
Despite the significant health, social and economic costs of cigarette smoking, 17% of Ontarians still currently smoke. Use of smoking cessation pharmacotherapy such as Zyban (bupropion HCl) has been shown to double quit rates but such medications are under-utilized by smokers attempting to quit. It has been suggested that the high price of pharmacotherapy may act as a barrier to accessing such treatment.The main objective of this study is to evaluate the methods and effectiveness of providing smokers who want to quit with 8 weeks of free Zyban in combination with smoking cessation counselling through family health teams and community health centres across the province.

Hypothesis: Ontario smokers who receive 8-weeks of free bupropion in combination with brief counselling will have higher smoking cessation rates than the standard population cessation rates.

DETAILED DESCRIPTION:
Nicotine dependence, like other addictive disorders, can be characterized as a chronic, relapsing disease (Leshner, 1997). Although there is significant morbidity and mortality associated with this disorder, the majority of smokers are not treated adequately to the widely accepted goal of complete long-term abstinence from smoking. This may be due to the under-utilization of accepted pharmacotherapies for the treatment of tobacco dependence.

Bupropion (Zyban) Bupropion is the first line of non-nicotine-based pharmacotherapy for smoking cessation. Several large-scale clinical trials have shown bupropion to be an efficacious smoking cessation aid (Hurt et al., 1997; Jorenby et al., 1999; Ahluwalia et al., 2002). In one such study, a 44% abstinence rate was reported for seven weeks of treatment with bupropion at 300 mg/day, compared to 19% for placebo (Hurt et al, 1997). A recent meta-analysis has reported that bupropion monotherapy approximately doubles the rate of smoking cessation (OR 1.94) (Hughes et al, 2007).

Despite its efficacy, bupropion's mechanism of action is unclear. Attenuation of abstinence-associated increase in craving and withdrawal symptoms has been suggested as possible mechanisms of bupropion's effect on smoking behaviour in a few randomized clinical trials (Jorneby et al., 1999; Shiffman et al., 2000; Lerman et al., 2002; Durcan et al, 2002). However, these effects are not universally demonstrated (Hurt et al., 1997; Shiffman et al., 2000). Other possible bio-behavioral mechanisms have remained largely unexplored. Using positron emission tomography (PET) it has been shown that in contrast to untreated smokers, when bupropion-treated smokers were exposed to cigarette-related cues there was less metabolic activation in their anterior cingulate cortex, a region of the brain previously shown to be activated by cigarette cues (Brody et al., 2004;Brody et al., 2002).

STOP Study Background and Rationale

Treatment with pharmacotherapy such as nicotine replacement therapy (NRT) or Zyban is a safe and effective smoking cessation strategy that can double the chance of quitting successfully over the long-term (Cornuz, 2007). However, research has shown that most smokers who are interested in quitting do not use pharmacotherapy to aid in their quit attempt. Misconceptions about the harmful effects of nicotine are a strong barrier to the use of pharmacotherapy. The cost of pharmacotherapy may also be a significant contributor to the under-utilization of smoking cessation aids such as NRT and Zyban. Karnath (2001) suggested that the high cost of successful pharmacotherapy treatment for smoking cessation may be a barrier for some individuals. Moreover, Cokkinides et al (2005) reported that smokers with private insurance were more likely to use smoking cessation pharmacotherapies than smokers without insurance. The addition of free NRT to a group behavioural cessation program substantiated these claims by showing an increase in quit rates from 38% to 65% (Alberg et al, 2004). These studies suggest that economic barriers may prevent smokers from using pharmacotherapy in their attempts to quit smoking.

The study proposed herein will introduce free bupropion as another treatment option for smoking cessation for Ontario smokers. Community Health Centres and Aboriginal Health Access Centres are interdisciplinary health models that are able to help individuals who would otherwise be prevented from accessing health services due to social and geographic barriers. As they aim to eliminate these other barriers and consequently control for them, they are an ideal health model for determining whether eliminating the economic barriers of smoking cessation improves smoking cessation rates. Family Health Teams are more recent health models that provide integrated and interdisciplinary primary health care. Since they are able to treat large and diverse populations, they are an ideal health model for accessing Ontario smokers.

Objectives

1. To evaluate the effectiveness of 8-weeks of free bupropion in combination with brief counselling through family health teams, community health centres and aboriginal health access centres in Ontario for smoking cessation.

ELIGIBILITY:
Inclusion Criteria:

* Ontario resident
* 18 years of age or older
* Current daily cigarette smoker who smokes 10 or more cigarettes per day and has smoked > 100 cigarettes in their lifetime
* Want to quit smoking cigarettes within 30 days of assessment
* Willingness and capacity to give written informed consent and to comply with study protocol

Exclusion Criteria:

* Enrollment in any of the STOP Study NRT models in the past 6 months
* Currently receiving Wellbutrin SR or any medication containing bupropion hydrochloride
* Current seizure disorder or history of seizures
* Current or prior diagnosis of bulimia or anorexia nervosa
* Current diagnosis of bipolar disorder
* History of head trauma
* Allergy or sensitivity to Zyban, Wellbutrin or bupropion
* Undergoing abrupt withdrawal from alcohol, benzodiazepines or other sedatives
* Currently taking monoamine oxidase (MAO) inhibitors, or thioridazine
* Pregnant or breastfeeding or at risk of becoming pregnant
* Central nervous system (CNS) tumor
* Severe hepatic impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 454 (Actual)
Dates: Start 2009-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Selby, MD, MHSc, Principal Investigator — Centre for Addiction and Mental Health
Locations (24):
- Canada (24):
  - The Youth Centre, Ajax, Ontario
  - Cottage Country Family Health Team, Bracebridge, Ontario
  - Bramalea Community Health Centre, Brampton, Ontario
  - Aberdeen Downtown Nurse Practitioner Clinic, Brantford, Ontario
  - Beausoleil Family Health Centre, Christian Island, Ontario
  - Georgian Bay Family Health Team, Collingwood, Ontario
  - North Renfrew Family Health Team, Deep River, Ontario
  - Elliot Lake Family Health Team, Elliot Lake, Ontario
  - Englehart & District Family Health Team, Englehart, Ontario
  - Stonegate Community Health Centre, Etobicoke, Ontario
  - Haliburton Highlands Family Health Team, Haliburton, Ontario
  - Algonquin Family Health Team, Huntsville, Ontario
  - Mary Beglund Community Health Centre, Ignace, Ontario
  - NorWest Community Health Centre, Longlac, Ontario
  - Summerville Family Health Team, Mississauga, Ontario
  - Mount Forest Family Health Team, Mount Forest, Ontario
  - Dufferin Area Family Health Team, Orangeville, Ontario
  - Somerset West Community Health Centre, Ottawa, Ontario
  - PrimaCare Community Family Health Team, Paris, Ontario
  - West Durham Family Health Team, Pickering, Ontario
  - Prince Edward Family Health Team, Picton, Ontario
  - Stratford Family Health Team, Stratford, Ontario
  - NorWest Community Health Centre, Thunder Bay, Ontario
  - Sandwich Community Health Centre, Windsor, Ontario

IPD SHARING:
Plan to Share IPD: No
No plan to share data

REFERENCES:
- [Background] Alberg AJ, Stashefsky Margalit R, Burke A, Rasch KA, Stewart N, Kline JA, Ernst PA, Avey A, Hoffman SC. The influence of offering free transdermal nicotine patches on quit rates in a local health department's smoking cessation program. Addict Behav. 2004 Dec;29(9):1763-78. doi: 10.1016/j.addbeh.2004.04.007. PMID 15530720
- [Background] Ahluwalia JS, Harris KJ, Catley D, Okuyemi KS, Mayo MS. Sustained-release bupropion for smoking cessation in African Americans: a randomized controlled trial. JAMA. 2002 Jul 24-31;288(4):468-74. doi: 10.1001/jama.288.4.468. PMID 12132977
- [Background] Brody AL, Mandelkern MA, London ED, Childress AR, Lee GS, Bota RG, Ho ML, Saxena S, Baxter LR Jr, Madsen D, Jarvik ME. Brain metabolic changes during cigarette craving. Arch Gen Psychiatry. 2002 Dec;59(12):1162-72. doi: 10.1001/archpsyc.59.12.1162. PMID 12470133
- [Background] Brody AL, Mandelkern MA, Lee G, Smith E, Sadeghi M, Saxena S, Jarvik ME, London ED. Attenuation of cue-induced cigarette craving and anterior cingulate cortex activation in bupropion-treated smokers: a preliminary study. Psychiatry Res. 2004 Apr 30;130(3):269-81. doi: 10.1016/j.pscychresns.2003.12.006. PMID 15135160
- [Background] Cokkinides VE, Ward E, Jemal A, Thun MJ. Under-use of smoking-cessation treatments: results from the National Health Interview Survey, 2000. Am J Prev Med. 2005 Jan;28(1):119-22. doi: 10.1016/j.amepre.2004.09.007. PMID 15626567
- [Background] Durcan MJ, Deener G, White J, Johnston JA, Gonzales D, Niaura R, Rigotti N, Sachs DP. The effect of bupropion sustained-release on cigarette craving after smoking cessation. Clin Ther. 2002 Apr;24(4):540-51. doi: 10.1016/s0149-2918(02)85130-x. PMID 12017399
- [Background] Hughes JR, Stead LF, Lancaster T. Antidepressants for smoking cessation. Cochrane Database Syst Rev. 2000;(4):CD000031. doi: 10.1002/14651858.CD000031. PMID 11034670
- [Background] Hurt RD, Sachs DP, Glover ED, Offord KP, Johnston JA, Dale LC, Khayrallah MA, Schroeder DR, Glover PN, Sullivan CR, Croghan IT, Sullivan PM. A comparison of sustained-release bupropion and placebo for smoking cessation. N Engl J Med. 1997 Oct 23;337(17):1195-202. doi: 10.1056/NEJM199710233371703. PMID 9337378
- [Background] Jorenby DE, Leischow SJ, Nides MA, Rennard SI, Johnston JA, Hughes AR, Smith SS, Muramoto ML, Daughton DM, Doan K, Fiore MC, Baker TB. A controlled trial of sustained-release bupropion, a nicotine patch, or both for smoking cessation. N Engl J Med. 1999 Mar 4;340(9):685-91. doi: 10.1056/NEJM199903043400903. PMID 10053177
- [Background] Leshner AI. Addiction is a brain disease, and it matters. Science. 1997 Oct 3;278(5335):45-7. doi: 10.1126/science.278.5335.45. PMID 9311924
- [Background] Lerman C, Roth D, Kaufmann V, Audrain J, Hawk L, Liu A, Niaura R, Epstein L. Mediating mechanisms for the impact of bupropion in smoking cessation treatment. Drug Alcohol Depend. 2002 Jul 1;67(2):219-23. doi: 10.1016/s0376-8716(02)00067-4. PMID 12095672
- [Background] Shiffman S, Johnston JA, Khayrallah M, Elash CA, Gwaltney CJ, Paty JA, Gnys M, Evoniuk G, DeVeaugh-Geiss J. The effect of bupropion on nicotine craving and withdrawal. Psychopharmacology (Berl). 2000 Jan;148(1):33-40. doi: 10.1007/s002130050022. PMID 10663415
- See also: Click here for more information about the study: STOP Study: Effectiveness of Zyban in a Clinical Population — http://www.stopstudy.ca
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching hospital, fully affiliated with the University of Toronto, and a PAHO/WHO Collaborating Centre. — http://www.camh.net/research

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bupropion HCl
Started | 454
Completed | 215
Not Completed | 239

BASELINE CHARACTERISTICS:
Population: Ontario smokers who are interested in quitting smoking.
Groups:
- Buproprion & Behavioural Support: 8 weeks of buproprion-SR + brief counselling for smoking cessation
Arm/Group | Buproprion & Behavioural Support
Number analyzed (Participants) | 454
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 415
  >=65 years | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.5 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 243
  Male | 211
Education level attained [Number; unit: participants] — highest level of education attained
  participants
    up to highschool | 238
    Post secondary | 207
    missing | 9
Employment [Number; unit: participants]
  Employed | 221
  Not employed | 229
  missing | 4
Income category [Number; unit: participants]
  up to $40,000 | 261
  more than $40,000 | 106
  missing | 87
Cigarettes per day (cpd) [Mean (Standard Deviation); unit: # cigarettes smoked per day] — # cigarettes smoked per day
  # cigarettes smoked per day | 20.5 (9.0)
Age first smoked [Mean (Standard Deviation); unit: years] | 14.1 (3.7)
Age smoked daily [Mean (Standard Deviation); unit: years] | 16.4 (4.3)
Time to first morning cigarette [Number; unit: participants]
  15 minutes or less | 306
  more than 15 minutes | 144
  missing | 4
# quit attempts in the past [Number; unit: participants]
  0 - 2 quit attempts | 181
  3 or more quit attempts | 225
  missing | 48
Importance of quitting smoking [Mean (Standard Deviation); unit: units on a scale] — scale of importance of quitting (1 to 10)
  1 - least important 10- most important
  units on a scale | 9.2 (1.3)
Confidence in quitting smoking [Mean (Standard Deviation); unit: units on a scale] — Confidence in quitting smoking
  1- very little confidence 10- very confident
  units on a scale | 7.6 (2.0)
Ever had a psychiatric diagnosis [Number; unit: participants]
  No | 309
  Yes | 145

OUTCOME MEASURES:

1. Primary Outcome: 7-day Point Prevalence of Smoking Abstinence
Description: Number of participants who report "Not Smoking (not even a puff) in past 7 days" when asked at week 8
Time Frame: End of Treatment (8 weeks after Zyban start date)
Population: Participants who completed survey 8 weeks after Zyban start date
Measure: Number; unit: participants
Groups:
- Nicotine Replacement & Behavioural Support: Nicotine Replacement Therapy: Transdermal nicotine patch, nicotine gum, nicotine inhaler, nicotine lozenge
  & Smoking cessation counselling-relapse prevention strategies.
Arm/Group | Nicotine Replacement & Behavioural Support
Number analyzed (Participants) | 215
participants
  Still smoking | 109
  Quit smoking | 106

2. Secondary Outcome: Serious Quit Attempt (at Least 24 Hours of Abstinence)
Description: Number of participants who report a serious quit attempt at End of treatment
Time Frame: End of Treatment (8 weeks after Zyban start date)
Population: This secondary outcome was not collected at 8 week followup.
Groups:
- Bupropion HCl and Counselling: Bupropion HCl Up to 8 week of bupropion SR (150mg BID) + counseling.
Arm/Group | Bupropion HCl and Counselling
Number analyzed (Participants) | 0

3. Secondary Outcome: 7-day Point Prevalence of Smoking Abstinence
Description: Number of participants who report "Not Smoking (not even a puff) in past 7 days" when asked 6 months after Zyban start date
Time Frame: 6 months after Zyban start date
Population: Number of participants who completed 6 month post treatment survey
Measure: Count of Participants; unit: Participants
Arm/Group | Buproprion & Behavioural Support
Number analyzed (Participants) | 448
Participants
  Smoked in past 7 days | 320
  Did not smoke in past 7 days | 128

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Bupropion HCl
Serious Adverse Events (participants affected / at risk) | 8/454
Other Adverse Events (participants affected / at risk) | 0/454
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bupropion HCl (N=454)
head injury (Injury, poisoning and procedural complications) | 1 (1) — Participant fell and hospitalized for head injury
wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) — ER visit for wheezing
Mental Health issues (Psychiatric disorders) | 2 (2) — ER visit for mental health issues
Chest pain (Cardiac disorders) | 1 (1) — ER visit for Chest pain
Pancreatitis (Gastrointestinal disorders) | 1 (1) — ER visit for Pancreatitis
Loss of consciousess (Nervous system disorders) | 2 (2) — Loss of consciousness

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No